CLINICAL TRIAL: NCT05338021
Title: Serum and Wound Vancomycin Levels Following Intrawound Administration in Primary Total Knee Arthroplasty
Brief Title: Intrawound Administration of Vancomycin in TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Xiang Shuai, MD, Principal Investigator, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AHQingdao VancoTKA
Record Dates: First submitted 2022-04-11; First posted 2022-04-20 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrawound Administration of Vancomycin (Experimental): After closure of the arthrotomy, 1 g of vancomycin powder suspended in 30ml of normal saline was injected directly into the joint with an 18-gauge needle. Then 20ml of normal saline was injected directly into the joint.
  Interventions: Procedure: Intrawound administration of vancomycin after closure of the arthrotomy
- Intrawound Administration of Vancomycin combined with epsilon-aminocaproic acid (EACA) (Experimental): After closure of the arthrotomy, 1 g of vancomycin powder suspended in 30ml of normal saline was injected directly into the joint with an 18-gauge needle. Then 4g (20ml) of epsilon-aminocaproic acid (EACA) was injected directly into the joint.
  Interventions: Procedure: Intrawound administration of vancomycin after closure of the arthrotomy

INTERVENTIONS:
Procedure: Intrawound administration of vancomycin after closure of the arthrotomy — After closure of the arthrotomy, 1 g of vancomycin powder suspended in 30ml of normal saline was injected directly into the joint with an 18-gauge needle.

SUMMARY:
The purpose of this study is to determine the intra-articular and serum levels of vancomycin over the first 24 hours postoperatively after intra-articular administration of a standard dose of vancomycin in primary total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50 and 80
2. Total knee arthroplasty for primary osteoarthritis. Primary diagnosis of knee osteoarthritis

Exclusion Criteria:

1. Diminished mental capacity
2. Vancomycin allergy
3. Chronic kidney disease stage III and stage IV

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Intra-articular vancomycin concentration | 2 hours, 8 hours and 24 hours postoperatively
Serum vancomycin concentration | 2 hours, 8 hours and 24 hours postoperatively
Renal function | Postoperative Day 1 and Day 3
  blood urea nitrogen (BUN), creatinine (Cr), GFR
Blood loss | Postoperative Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Xiang, M.D., Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The affiliated hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: After completing this trial.

REFERENCES:
- [Derived] Li X, Lai J, Yang X, Xu H, Xiang S. Intra-articular injection of vancomycin after arthrotomy closure following gentamicin-impregnated bone cementation in primary total knee arthroplasty provides a high intra-articular concentration while avoiding systemic toxicity: a prospective study. J Orthop Surg Res. 2024 Dec 19;19(1):856. doi: 10.1186/s13018-024-05357-9. PMID 39702402